CLINICAL TRIAL: NCT02104011
Title: Treatment of Renal Angiomyolipomas in Tuberous Sclerosis by Beta-blockers: Pilot Trial
Brief Title: Treatment of Renal Angiomyolipomas in Tuberous Sclerosis by Beta-blockers
Acronym: STBETA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2011/35
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Renal Angiomyolipomas; Tuberous Sclerosis
Keywords: Angiomyolipomas in tuberous sclerosis; Beta-blockers; Anti-angiogenic therapies
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient (Experimental)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol

SUMMARY:
Treatment of angiomyolipomas is based on invasive techniques such as surgery or embolization. Development of anti-angiogenic therapies is a major and growing field of research in hypervascularized tumors. Angiomyolipomas have been shown to regress after prolonged treatment with mTOR inhibitors (Sirolimus), but with a large proportion of secondary effects. We showed recently that beta-blockers were able to induce regression of infantile hemagiomas. Consequently, we looked for and found, histologically, in a few cases of angiomyolipomas the presence of beta2 receptors.

The aim of the study is to estimate if beta-blockers could induce regression or stabilization of renal angiomyolipomas in tuberous sclerosis in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Tuberous sclerosis patients with one or several angiomyolipomas of a size of at least 4 cms.

Exclusion Criteria:

* Patients whom CT or MR scan shows one or several intra-lesional aneurisms requiring a preventive embolization.
* Patients with a retroperitoneal hemorragic complication requiring a preventive embolization.
* Patients whom biopsy will show an adenocarcinoma, hypertension non controlled, renal failure and severe liver.
* Diabetic subjects insufficiently controlled.
* Beta-blockers contra-indication.
* Psychosis, severe mental disorder.
* Patient already treated with beta-blockers or mTOR inhibitors.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Evolution of angiomyolipomas volume | 6 months and 1 year after inclusion
  Stabilization or even regression of angiomyolipomas volume after 6 months and 1 year of treatment with a quantification of the vascular component.

SECONDARY OUTCOMES:
Renal function evolution | 6 months and 1 year after inclusion
  Improvement of renal function after 6 months and 1 year of treatment
Effect on the potential haemorraghic transformation | 6 months and 1 year after inclusion
  Haemorraghic transformation of angiomyolipomas is diagnosed by Scanner or MRI.
Improvement of the quality of life | 6 months and 1 year after inclusion.
  Th evolution of the quality of life is assessed by an EVA scale and by QOL scale.
Effect on face angiofibromas | 6 months and 1 year after inclusion
  Evolution of the face angiofibromas by a dermatologic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Claire RIGOTHIER, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Nephrology department, Bordeaux, France